CLINICAL TRIAL: NCT00554034
Title: The Effect of Herbal Extracts on Inflammatory Enzymes in the Gingiva: a Dose Finding Study.
Brief Title: Effect of Herbal Extracts on Gingival Inflammation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Menachem Oberbaum, MD, Shaare Zedek Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol C-4
Record Dates: First submitted 2007-10-15; First posted 2007-11-06 (Estimated); Last update posted 2010-12-21 (Estimated); Status verified 2009-04

CONDITIONS: Gingivitis
Keywords: gingivitis, localized treatment
MeSH Terms: conditions — Gingivitis

INTERVENTIONS:
Drug: periopatch — Patients enrolled in the study will be given 1, 2, 3 or 4 patches in a cycle by the order they enter the study.

SUMMARY:
The purpose of this study is to determine the minimal number of patches needed to get an effective response. Patients enrolled in the study will be given 1, 2, 3 or 4 patches in a cycle by the order they enter the study. After the first 20 patients [5 cycles], the effect of the number of patches will be tested. If there is no distinct reduction of beta glucuronidase in the GCF or of gingival index at the tested sites, more patients will be enrolled. Patients will be added one cycle at a time with results being tested and analyzed. The enrollemnts of patients will stop when a dose response will be noticed or 15 cycles have been reached.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 -75.
2. Severe localized gingival inflammation [GI index 2 or greater

Exclusion Criteria:

1. Pregnancy or a wish to become pregnant during the study.
2. History of periodontal treatment within the last month.
3. Antibiotic treatment within the last month
4. Use of any antimicrobial mouthrinse within the last month.
5. Participation in another trial one month prior to the study.
6. Inability to behave compliant to the trial protocol by not placing all the patches given, or attending scheduled appointments.
7. Systemic Disease.
8. Patients using salicylate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-11; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To determine the correct dosing of the herbal Patch [THPP] | 3 months

SECONDARY OUTCOMES:
To demonstarte the safety of THPP on the gingival tissue and in the oral cavity | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Menachem Oberbaum, M.D., Principal Investigator — Shaare Zedek Medical Center, Jerusalem, Israel
Locations (1):
- Jerusalem Perio Center, Jerusalem, Israel